CLINICAL TRIAL: NCT02322580
Title: Intermittent Versus Continuous Treatment: an Observational Monocentric Study Investigating the Association Between Trough Levels of Enbrel and Therapy Regimen
Brief Title: An Observational Monocentric Study Investigating the Association Between Trough Serum Levels of Etanercept, Antibodies Towards Etanercept and Its Effectiveness in Psoriasis Patients
Acronym: DERM
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: S56818
Record Dates: First submitted 2014-12-11; First posted 2014-12-23 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-05

CONDITIONS: Psoriasis
Keywords: anti-TNF; therapeutic drug monitoring; immunogenicity
MeSH Terms: conditions — Psoriasis | interventions — Etanercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Psoriasis patients who receive Enbrel® therapy
  Interventions: Drug: etanercept

INTERVENTIONS:
Drug: etanercept
  Other Names: Enbrel®

SUMMARY:
The purpose of this study is to investigate the association between trough serum levels of etanercept, antibodies towards etanercept and its effectiveness in psoriasis patients.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 years on, male or female
* Established diagnosis of psoriasis
* Etanercept either on monotherapy or in combination with acitretin (Neotigason®), given according to the current EU SmPC including the safety measures.
* Patients who give informed consent for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Psoriasis patients who receive Enbrel® therapy according to the current EU Summary of Product Characteristics (SmPC)
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2015-01; Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
trough serum etanercept concentration | one year
anti-etanercept serum concentration | one year